CLINICAL TRIAL: NCT06257719
Title: Clinical Characteristics of Lymphatic Malformations: An Observational Study
Brief Title: Clinical Characteristics of Lymphatic Malformations
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Principal Investigator, West China Hospital
Other Study IDs: 2024-127
Record Dates: First submitted 2024-01-16; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Lymphatic Malformation; Lymphangioma
Keywords: Lymphatic Malformation; Abdominal site; Preoperative complications; Resection; Mesentery; Acute abdomen
MeSH Terms: conditions — Lymphatic Abnormalities; Lymphangioma; Abdomen, Acute | interventions — Surgical Procedures, Operative; Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paediatric group: The investigators defined participants under 14 years old as the paediatric group.
  Interventions: Other: Compare the epidemiological characteristics, clinical presentations, surgical treatments and risk factors for preoperative complications of ALMs between paediatric and adult participants.
- Adult group: The investigators defined participants over 14 years old as the adult group.
  Interventions: Other: Compare the epidemiological characteristics, clinical presentations, surgical treatments and risk factors for preoperative complications of ALMs between paediatric and adult participants.

INTERVENTIONS:
Other: Compare the epidemiological characteristics, clinical presentations, surgical treatments and risk factors for preoperative complications of ALMs between paediatric and adult participants. — Compare the epidemiological characteristics, clinical presentations, surgical treatments and risk factors for preoperative complications of ALMs between paediatric and adult participants.

SUMMARY:
The primary purpose of this study is to retrospectively identify the clinical characteristics of abdominal lymphatic malformations (ALMs) in our single center in China. The second objective of this study is to retrospectively compare the epidemiological features, clinical presentations, cyst properties, surgical treatments, and risk factors for preoperative complications of ALMs between paediatric participants and adult participants.

DETAILED DESCRIPTION:
Lymphatic malformations (LMs) are vascular anomalies that arise from abnormal embryonic development of the lymphatic system and can present as dilated lymphatic channels or cysts lined by lymphatic endothelial cells. Abdominal lymphatic malformations (ALMs) are rare entities that account for fewer than 10% of LMs and may occur not only in the tissues or organs in the abdominal cavity, such as the mesentery, spleen and pancreas but also in the retroperitoneal space. ALMs can manifest as an infection, chronic abdominal discomfort, acute abdomen, or fatal disease.

ELIGIBILITY:
Inclusion Criteria:

* The investigators enrolled participants who were pathologically diagnosed with lymphangioma or lymphatic malformations in the abdominal cavity (i.e., abdominal lymphatic malformations) from January 2009 to December 2022 at our institution.

Exclusion Criteria:

* The investigators excluded participants without a pathological diagnosis of abdominal lymphatic malformations through resection specimens and those with pathological confirmation of other diseases, as well as patients with complex lymphatic anomalies.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In this study, The investigators retrospectively collected and compared the data related to the preoperative information, intraoperative findings and postoperative pathological analysis of the enrolled abdominal lymphatic malformations for paediatric and adult participants.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
The location of abdominal lymphatic malformations in participants | From 2009.1 to 2022.12
  Location included mesentery, retroperitoneum, omentum, spleen, etc.
The morphologic subtypes of abdominal lymphatic malformations in participants | From 2009.1 to 2022.12
  Morphologic subtypes included macrocystic, microcystic and mixed type.
The presentations at diagnosis of abdominal lymphatic malformations in participants | From 2009.1 to 2022.12
  Presentations at diagnosis included chronic pain, acute abdominal disease and incidental health checkup.
The largest diameter of abdominal lymphatic malformations in participants | From 2009.1 to 2022.12
  Largest diameter in centimeters was mainly measured by intraoperative detections.
The preoperative complications of abdominal lymphatic malformations in participants | From 2009.1 to 2022.12
  Preoperative complications included intestinal volvulus, haemorrhage, infection, rupture and compression.

SECONDARY OUTCOMES:
The incidence of abdominal lymphatic malformations in paediatric and adult group | From 2009.1 to 2022.12
  Incidence of abdominal lymphatic malformations in paediatric and adult group was retrospectively compared.
The number of female patients with abdominal lymphatic malformations in paediatric and adult group | From 2009.1 to 2022.12
  Number of female patients with abdominal lymphatic malformations in paediatric and adult group was retrospectively compared.
The rate of abdominal lymphatic malformations with acute abdomen in paediatric and adult group | From 2009.1 to 2022.12
  Rate of abdominal lymphatic malformations with acute abdomen in paediatric and adult group was retrospectively compared.
The rate of abdominal lymphatic malformations located in mesentery for paediatric and adult group | From 2009.1 to 2022.12
  Rate of abdominal lymphatic malformations located in mesentery for paediatric and adult group was retrospectively compared.
The risk factors of preoperative complications of abdominal lymphatic malformations for paediatric and adult group. | From 2009.1 to 2022.12
  Risk factors of preoperative complications of abdominal lymphatic malformations for paediatric and adult group was retrospectively compared.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ji, Ph.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No